CLINICAL TRIAL: NCT04645056
Title: The Impact of Post-thyroidectomy Neck Stretching Exercises on Improving Short Term Quality of Life: A Randomized Prospective Clinical Trial
Brief Title: The Impact of Post-thyroidectomy Neck Stretching Exercises on Improving Short Term Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Rehabilitation thyroidectomy
Record Dates: First submitted 2020-07-01; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-04

CONDITIONS: Thyroidectomy
Keywords: Rehabilitation; Stretching; Otolaryngology; Quality of Life; Musculoskeletal Pain; Neck Pain; Voice Quality
MeSH Terms: conditions — Musculoskeletal Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: Patients will be recruited for this randomized controlled clinical study the day after surgery. Participants are randomized into two groups using a randomization scheme according to whether the surgery is performed in a week with an even or uneven number (e.g. week number 42 or 43 within a given year). A designated person with no impact on the decision of surgical procedure will handle the randomization and recruitment (the project owner).
  The patients are randomized to either intervention with nine specific and carefully selected neck stretching exercises or to the control group without any intervention.
  Before discharge, both groups are instructed to perform either stretching exercises or to no intervention, respectively, the four postoperative weeks. A follow-up phone call will be made approximately one week after discharge to ensure patient adherence.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): a. Intervention Group: Neck stretching and movement
  The patient starts the stretching exercises the morning after surgery with instructions from a trained professional at the department. The patient is informed that the stretching exercises will not affect the surgical wound. The patient is instructed in performing five repetitions of each of the following nine exercises three times each day in four weeks:
  1. Relax shoulders and neck sufficiently
  2. Look down - Stretching and movement
  3. Look to each side - movement
  4. Lower the head to each side - stretching
  5. Lower the head diagonally to each side - stretching
  6. Small nod movements
  7. Lift the shoulders - movement
  8. Roll the shoulders - movement
  9. Lift the arms - movement
  The first stretching session is observed by the instructor who gives feedback and correct the exercises, if necessary. Furthermore, the patient is given a training brochure.
  Interventions: Other: Stretching and Mobility exercises for neck and shoulder
- Control group (No Intervention): b. Control group The patients in the control group are not instructed in any intervention but are answering completely similar questionnaires as the intervention group.

INTERVENTIONS:
Other: Stretching and Mobility exercises for neck and shoulder — 9 specific stretching and mobility exercises performed 3 times every day the first 4 weeks after surgery.
  Arms: Intervention group

SUMMARY:
The project deals with patients undergoing surgery in the neck due to benign tumor in the thyroid gland in order to remove pressure symptoms.

The background of the project is a recent series of studies (Sorensen, Watt et al. 2017) (Sorensen, Watt et al. 2017), showing that patients are very adversely affected by a reduced voice function and pain the neck/shoulders in the first weeks and months after the operation. In general, the patients quality of life is impaired in this period. Due to this, it is relevant to seek ways to reduce the discomfort symptoms after the operation by performing simple and specific chosen stretching exercises for the muscles in the neck and shoulders.

The patients in the project are randomly divided into two groups, and both groups are answering questionnaires after 1,2, 4 weeks and after 3 months regarding their short time quality of life focusing on voice function and pain in the neck and shoulders. The patients in the intervention group are instructed in stretching and mobility exercises for neck and shoulder starting the day after surgery and they are supposed to perform them every day in four weeks after surgery. The control group are not performing these exercises and are not informed that there concurrently is an intervention going on. In this way the questionnaires can be compared in the end.

The hypothesis is that short time quality of life including voice function and pain the neck and shoulder can be improved for this group of patients with these specific stretching and mobility exercises. The project is of great clinical relevance and can in case of confirmed hypothesis be applied in clinical practice immediately benefitting the patients undergoing surgery.

DETAILED DESCRIPTION:
PROJECT DESCRIPTION

Background/introduction:

Removing all or part of the thyroid gland by surgery, has routinely been used for more than 100 years for the treatment of patients with benign as well as malignant thyroid disease. It is generally accepted that quality of life is improved three-to-six months after surgery (Mishra, Sabaretnam et al. 2013) (Sorensen, Watt et al. 2017) (Watt, Cramon et al. 2014). However, in the days and weeks following thyroid surgery, patients often experience muscle pain and stiffness of the neck and shoulders (Yuuki Takumara 2005). In addition, 2-4 weeks postoperatively voice discomfort symptoms can be pronounced, and although short-termed and passing, patients experience a decreased quality of life (Sorensen, Printz et al. 2019) (Vicente, Solomon et al. 2014) (Ryu, Ryu et al. 2013). The accumulation of such symptoms in the weeks just after surgery may reduce quality of live significantly. Therefore, any rehabilitative interventions which may reduce discomfort are highly relevant.

A limited number of randomized trials have investigated the effect of early postoperative rehabilitative measures such as neck stretching. Rehabilitation with stretching exercises is found to reduce neck pain, neck stiffness, and the need for postoperative pain relief medication (Yuuki Takumara 2005) (Hatice Ayhan 2016). No study has examined the effect of neck stretching exercises on short term quality of life improvements in relation to voice function despite many of the neck muscles are used for voice production. The same goes for the impact of neck stretching exercises on short term quality of life improvements in relation to neck pain.

Objective/Purpose The objective is to examine the effect of neck stretching exercises performed shortly after hemi- and total thyroidectomy on short term quality of life in relation to subjective voice function and neck pain in the first four weeks after surgery.

Study population In-hospital patients with benign thyroid disease having undergone thyroid surgery at the Department of Otorhinolaryngology (ORL) - Head & Neck Surgery, Odense University Hospital.

Study Design and patient recruitment Patients will be recruited for this randomized controlled clinical study the day after surgery. Participants are randomized into two groups using a randomization scheme according to whether the surgery is performed in a week with an even or uneven number (e.g. week number 42 or 43 within a given year). A designated person with no impact on the decision of surgical procedure will handle the randomization and recruitment (the project owner).

The patients are randomized to either intervention with nine specific and carefully selected neck stretching and mobility exercises or to the control group without any intervention.

Before discharge, both groups are instructed to perform either stretching exercises or to no intervention, respectively, the four postoperative weeks. A follow-up phone call will be made approximately one week after discharge to ensure patient adherence.

Methods The effect will be examined for both the intervention group and control group through an electronic questionnaire comprising three parts (see below) with focus on short term quality of life, subjective voice function, and neck pain, respectively. A baseline status will be made by the patient at enrollment on the first postoperative day, by recalling the four weeks prior to surgery.

The questionnaires will be answered a total of three times during the 4 weeks postoperative period. The questionnaires will be delivered by a secure email system one week, two weeks, four weeks and three months after surgery. Futhermore, every patient in both groups will take a blood sample four weeks postoperative to examine the level of TSH (thyroid-stimulating hormone).

Randomization groups (see "arms")

1. Intervention Group: Neck stretching
2. Control group: No intervention

Questionnaires

1. Thyroid-Related Patient-Reported Outcome (ThyPRO-39) ThyPRO is a patient-reported outcome covering Quality of Life symptoms specifically validated for patients with benign thyroid diseases, including patients undergoing thyroidectomy. The ThyPRO consists of 39 items and is rated by the patient on a Likert scale from 0-4 with 0 = no symptoms/problems and 4 = Severe symptoms/problems (Watt, Bjorner et al. 2015).
2. Numeric Rating Scale (NRS Pain Score) The Numerical Rating Scale is a pain assessment tool by which the patient is asked to rate their pain on a scale between 0 and 10 (0 represents "no pain" and 10 represents "the worst pain ever possible") (Haefeli and Elfering 2006)
3. Voice handicap Index 10 The Voice Handicap Index-10 (VHI-10) is a scale designed to focus on the patients' self-perception of their voice disorders. The VHI-10 is a list of ten statements, each of which is evaluated by the patient on a five-point Likert like scale (0-4 points) in relation to the frequency of their experienced voice symptoms (never, almost never, sometimes, almost always, always) (Michael S. Benninger 1998).
4. European Quality Of Life (EQ-5D) The EQ-5D is a standardized non-disease specific instrument to describe and value health-related quality of life. The questionnaire consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Futhermore, it ends with a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine from 0 to 100. (Foundation 2020, June 09)

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing either hemi- or total thyroidectomy for a benign thyroid disease

Exclusion Criteria:

* Pre-operative recurrent laryngeal nerve palsy
* Pre-operative voice disorder requiring treatment by surgery or speech language pathology
* Previous neck surgery including thyroid surgery
* Patients under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Short time quality of life (QoL) | Short time QoL 1 week after surgery
  Short time quality of life including voice quality and pain in neck and shoulders measured in specific questionnaires answered before and 4 times after surgery (2 weeks before, 1,2,4 weeks and 3 months after surgery).
Short time quality of life (QoL) | Short time QoL 2 weeks after surgery
  Short time quality of life including voice quality and pain in neck and shoulders measured in specific questionnaires answered before and 4 times after surgery (2 weeks before, 1,2,4 weeks and 3 months after surgery).
Short time quality of life (QoL) | Short time QoL 4 weeks after surgery
  Short time quality of life including voice quality and pain in neck and shoulders measured in specific questionnaires answered before and 4 times after surgery (2 weeks before, 1,2,4 weeks and 3 months after surgery).
Short time quality of life (QoL) | Short time QoL three months after surgery
  Short time quality of life including voice quality and pain in neck and shoulders measured in specific questionnaires answered before and 4 times after surgery (2 weeks before, 1,2,4 weeks and 3 months after surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Godballe, Doctor, Study Director — Department of ENT Head & Neck Surgery, Odense University Hospital, Denmark
Locations (1):
- Department of ENT Head & Neck Surgery, Odense University Hospital, Denmark, Odense C, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Ayhan H, Tastan S, Iyigun E, Ozturk E, Yildiz R, Gorgulu S. The Effectiveness of Neck Stretching Exercises Following Total Thyroidectomy on Reducing Neck Pain and Disability: A Randomized Controlled Trial. Worldviews Evid Based Nurs. 2016 Jun;13(3):224-31. doi: 10.1111/wvn.12136. Epub 2016 Jan 15. PMID 26773539
- [Background] Benninger MS, Ahuja AS, Gardner G, Grywalski C. Assessing outcomes for dysphonic patients. J Voice. 1998 Dec;12(4):540-50. doi: 10.1016/s0892-1997(98)80063-5. PMID 9988041
- [Background] Mishra A, Sabaretnam M, Chand G, Agarwal G, Agarwal A, Verma AK, Mishra SK. Quality of life (QoL) in patients with benign thyroid goiters (pre- and post-thyroidectomy): a prospective study. World J Surg. 2013 Oct;37(10):2322-9. doi: 10.1007/s00268-013-2133-3. PMID 23838927
- [Background] Ryu J, Ryu YM, Jung YS, Kim SJ, Lee YJ, Lee EK, Kim SK, Kim TS, Kim TH, Lee CY, Park SY, Chung KW. Extent of thyroidectomy affects vocal and throat functions: a prospective observational study of lobectomy versus total thyroidectomy. Surgery. 2013 Sep;154(3):611-20. doi: 10.1016/j.surg.2013.03.011. Epub 2013 Aug 8. PMID 23932596
- [Background] Sorensen JR, Printz T, Iwarsson J, Grontved AM, Dossing H, Hegedus L, Bonnema SJ, Godballe C, Mehlum CS. The Impact of Post-thyroidectomy Paresis on Quality of Life in Patients with Nodular Thyroid Disease. Otolaryngol Head Neck Surg. 2019 Oct;161(4):589-597. doi: 10.1177/0194599819855379. Epub 2019 Jun 11. PMID 31184263
- [Background] Sorensen JR, Watt T, Cramon P, Dossing H, Hegedus L, Bonnema SJ, Godballe C. Quality of life after thyroidectomy in patients with nontoxic nodular goiter: A prospective cohort study. Head Neck. 2017 Nov;39(11):2232-2240. doi: 10.1002/hed.24886. Epub 2017 Sep 4. PMID 28872214
- [Background] Vicente DA, Solomon NP, Avital I, Henry LR, Howard RS, Helou LB, Coppit GL, Shriver CD, Buckenmaier CC, Libutti SK, Shaha AR, Stojadinovic A. Voice outcomes after total thyroidectomy, partial thyroidectomy, or non-neck surgery using a prospective multifactorial assessment. J Am Coll Surg. 2014 Jul;219(1):152-63. doi: 10.1016/j.jamcollsurg.2014.03.019. Epub 2014 Mar 18. PMID 24745621
- [Background] Watt T, Bjorner JB, Groenvold M, Cramon P, Winther KH, Hegedus L, Bonnema SJ, Rasmussen AK, Ware JE Jr, Feldt-Rasmussen U. Development of a Short Version of the Thyroid-Related Patient-Reported Outcome ThyPRO. Thyroid. 2015 Oct;25(10):1069-79. doi: 10.1089/thy.2015.0209. Epub 2015 Aug 26. PMID 26214034
- [Background] Watt T, Cramon P, Frendl DM, Ware JE Jr; ThyQoL Group. Assessing health-related quality of life in patients with benign non-toxic goitre. Best Pract Res Clin Endocrinol Metab. 2014 Aug;28(4):559-75. doi: 10.1016/j.beem.2014.01.009. Epub 2014 Jan 28. PMID 25047206
- [Background] Takamura Y, Miyauchi A, Tomoda C, Uruno T, Ito Y, Miya A, Kobayashi K, Matsuzuka F, Amino N, Kuma K. Stretching exercises to reduce symptoms of postoperative neck discomfort after thyroid surgery: prospective randomized study. World J Surg. 2005 Jun;29(6):775-9. doi: 10.1007/s00268-005-7722-3. PMID 16078129
- [Derived] Thorsen RT, Dossing H, Bonnema SJ, Brix TH, Godballe C, Sorensen JR. The Impact of Post-Thyroidectomy Neck Stretching Exercises on Neck Discomfort, Pressure Symptoms, Voice and Quality of Life: A Randomized Controlled Trial. World J Surg. 2022 Sep;46(9):2212-2222. doi: 10.1007/s00268-022-06610-0. Epub 2022 May 30. PMID 35637354